The Anti-Inflammatory Effects of Exercise and Peanut Consumption

PI: Richard P. Sloan, PhD

IRB# 7466

NCT03212144

May 25, 2018

## Statistical Analysis Plan

As this is only a pilot study, we plan simply to test change scores in inflammatory markers from laboratory session 1 to 2 and 3 to 4 for participants in the two arms. Specifically, change scores for the peanut intervention will be compared to change scores for the exercise intervention using a within-subject t-test.